CLINICAL TRIAL: NCT06044038
Title: Enhancing Functional Capacity and Body Composition of Individuals With Schizophrenia Through a Physical Exercise Intervention
Brief Title: Exercise Intervention for People With Schizophrenia (CREW)
Acronym: CREW
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Università degli Studi di Ferrara (Other)
Responsible Party: Principal Investigator, Mandini Simona, Professor, Università degli Studi di Ferrara
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CSB-23-02
Record Dates: First submitted 2023-09-05; First posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Physical activity; Mental disorder
MeSH Terms: conditions — Schizophrenia; Motor Activity; Mental Disorders | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physical activity group (Experimental): Participation in supervised activities such as walking or Nordic walking groups, gentle gymnastics, soccer, swimming, and volleyball. Each activity was scheduled twice a week.
  Interventions: Behavioral: Physical activity; Behavioral: Cognitive rehabilitation program
- Usual care group (Other): Participants in the control group attended weekly 90-minute cognitive rehabilitation sessions according to the usual care procedure in this type of population.
  Interventions: Behavioral: Cognitive rehabilitation program

INTERVENTIONS:
Behavioral: Physical activity — Bi-weekly supervised physical activity intervention
  Arms: Physical activity group
Behavioral: Cognitive rehabilitation program — weekly 90-minute session consisting of welcoming participants, reviewing tasks conducted in the last meeting, and assignment of new pen-and-pencil cognitive and metacognitive tasks.

SUMMARY:
The study aims to investigate the feasibility and adherence of long-term, moderate-intensity different types of physical activity programs for individuals with schizophrenia. Secondary outcomes are related to the control of non-communicable disease risk factors and the improvement of exercise capacity, body composition and cognitive function.

DETAILED DESCRIPTION:
Schizophrenia is a common public health issue that generates a social and economic burden. Individuals affected by schizophrenia experience severe and chronic levels of disability that derive from acute psychotic symptoms, as well as cognitive impairments for which available treatments offer only limited benefits. Moreover, their life expectancy is lower, and they have a higher prevalence of heart diseases risk factors such as obesity, dyslipidemia, smoking, hypertension, diabetes and physical inactivity than the general population. The World Health Organization and the European Mental Health Action Plan 2013-2020 acknowledge the role of physical activity in mental health and encourage the inclusion of lifestyle changes in education and treatment programs for people with mental illness, delivered in primary and secondary healthcare settings. The benefits of regular physical activity are well-recognized and are inversely associated with mortality risk and the incidence of many chronic diseases. Moreover, it plays a critical role in preserving and even improving cognitive function throughout the lifespan. However, people with schizophrenia tend to be less engaged in physical activity programs than the general population and report a range of barriers such as pain, side effects of medications and negative symptoms.

The purpose of this trial is to evaluate the efficacy of an exercise-based intervention program among people with schizophrenia.

All individuals with schizophrenia were screened for eligibility. After verifying inclusion and exclusion criteria and after eligibility is confirmed, written informed consent must be obtained prior to randomization. Baseline patient characteristics (i.e., demographics, medical history, laboratory test results) have been collected and recorded for further assessment. Randomization was performed during the inclusion visit (T1). Randomization will be performed centrally using an internet-based system. The identification number (ID) and the treatment allocation will be assigned by the randomization system. Patients were randomized to physical activity group or usual care by a 2:1 allocation. After the randomization, all participants underwent the same battery of tests and questionnaires according to the study protocol.

All patients were involved in the usual care cognitive program. It was held in weekly 90-minute sessions in a Psychiatric Rehabilitation Center of the Healthcare District of Ferrara. Specialized psychiatric therapists conduct this program with groups of 5-10 participants, based on a Cognitive Remediation model. Each session consists of welcoming participants, reviewing tasks conducted in the last meeting, and assignment of new pen-and-pencil cognitive and metacognitive tasks. Tasks include games and exercises (e.g., sudoku, crosswords), as well as discussions aimed at improving short- and long-term memory (i.e., repeating sequences of words and numbers), executive functions, and social cognition, with progressive adaptation of task difficulty. The total number of sessions is 50 for a duration of 12 months. In addition, the intervention arm was involved in a supervised exercise-based program. They could voluntarily participate in a variety of activities such as walking or Nordic walking groups, gentle gymnastics, soccer, swimming, and volleyball. Each activity was scheduled twice a week.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with schizophrenia for at least 1 year
* On antipsychotic medications with the same therapeutic regimen for at least 3 months before enrolment
* Free of symptomatic peripheral arterial occlusive disease and cardiovascular, pulmonary, neurological, metabolic, and orthopaedic disorders that could interfere with physical activity sessions

Exclusion Criteria:

* Recent modification of the therapeutic regimen
* Presence of symptomatic peripheral arterial occlusive disease and cardiovascular, pulmonary, neurological, metabolic, and orthopaedic disorders that could interfere with physical activity sessions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-12-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Peak Oxygen Uptake (VO2peak) | First assessment at the date of enrolment (baseline) and subsequently every six months until the date of the end of follow-up (up to 2 years)
  Measurement of cardiorespiratory fitness, reported as ml/kg/min and estimated through a moderate and perceptually regulated 1km treadmill walk test (1k-TWT) or through related short-forms (500m or 200m)
Body Mass Index (kg/m²) | First assessment at the date of enrolment (baseline) and subsequently every six months until the date of the end of follow-up (up to 2 years)
  Derived from the measurement of weight in kilograms and height in meters
Waist circumference (cm) | First assessment at the date of enrolment (baseline) and subsequently every six months until the date of the end of follow-up (up to 2 years)
  Measurement of waist circumference
Screen for Cognitive Impairment in Psychiatry (SCIP) | First assessment at the date of enrolment (baseline) and subsequently every six months until the date of the end of follow-up (up to 2 years)
  Values range from 0 to >100, higher scores mean a better outcome
Frontal Assessment Battery (FAB) | First assessment at the date of enrolment (baseline) and subsequently every six months until the date of the end of follow-up (up to 2 years)
  Values range from 0 to18, higher scores mean a better outcome

SECONDARY OUTCOMES:
Adherence | From date of enrollment until the date of the end of follow-up (up to 2 years)
  Number of physical activity sessions attended by the participants and the number of drop-outs

CONTACTS AND LOCATIONS:
Overall Officials: Gianni Mazzoni, Professor, Study Director — Università degli Studi di Ferrara; Simona Mandini, PhD, Principal Investigator — Università degli Studi di Ferrara
Locations (1):
- Center for Exercise Science and Sport, Ferrara, Italy

REFERENCES:
- [Result] Mandini S, Morelli M, Belvederi Murri M, Grassi L, Masotti S, Simani L, Zerbini V, Raisi A, Piva T, Grazzi G, Mazzoni G. Adherence to a guided walking program with amelioration of cognitive functions in subjects with schizophrenia even during COVID-19 pandemic. BMC Sports Sci Med Rehabil. 2022 Mar 25;14(1):48. doi: 10.1186/s13102-022-00440-2. PMID 35337370